CLINICAL TRIAL: NCT06547281
Title: Elderly Surgical Patients Multi-Infection Prediction: Machine Learning Model Development & Validation With SHAP Analysis
Brief Title: Machine Learning Prediction of Multiple Infections in Elderly Surgical Patients
Status: Completed | Type: Observational
Sponsor: Weidong Mi (Other)
Responsible Party: Sponsor-Investigator, Weidong Mi, Depatment of Anesthesiology, The First Medical Center, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: PLAGH-AOC-L03
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Infection; Geriatrics; Prediction
Keywords: the elderly; postoperative infection; machine learning; risk model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Utilizing machine learning techniques, investigators developed the geriatric infection assessment model, leveraging domestic databases to predict multiple postoperative infections in elderly patients. The model addresses the current gap in predictive tools tailored for elderly surgical patients in China, offering insights into both overall and specific infection risks.

DETAILED DESCRIPTION:
Backgrounds:

Postoperative infections are a leading cause of adverse perioperative outcomes, particularly for elderly patients. Given the varied diagnostic presentations of infection, there is a significant gap in the use of predictive tools to identify those at high risk of developing such complications.

Objective:

Investigators aimed at developing machine learning models to predict various postoperative infection risks in elderly patients, facilitating early detection and intervention.

Methods:

A retrospective analysis was conducted on 42,540 elderly patients who underwent non-cardiac surgery at the First Medical Center of the Chinese PLA General Hospital between January 2012 and August 2018, forming the Training set. From this, a 30% subset was randomly designated as the Test set. The models incorporated 51 variables including key infection-related factors. Three machine learning techniques-Logistic Regression (LR), Random Forest (RF), and Gradient Boosting Machines (GBM)-were utilized to develop predictive models for overall and specific postoperative infections, categorized according to the European Perioperative Clinical Outcome (EPCO) definitions. Model performance was gauged by metrics such as the Area Under the Receiver Operating Characteristic (ROC) Curve (AUC), accuracy, and precision. To enhance model interpretability, investigators employed the RF model's Variable Importance (VIMP) and Shapley Additive Explanations (SHAP) algorithm. For a demonstrable prediction of specific infection types, data of randomly selected 5 patients were fed into the model with the resulting probabilities depicted in a radar chart.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years;
2. Patients undergoing surgeries not involving local anesthesia.

Exclusion Criteria:

1. Patients undergoing neurosurgery or cardiac surgery;
2. Patients with preoperative infections (including pneumonia, SSIs, UTIs, and bloodstream infections).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Training set included 42,540 elderly patients treated at the First Medical Center of the Chinese PLA General Hospital (PLAGH) from January 2012 to August 2018.
Sampling Method: Non-Probability Sample
Enrollment: 42540 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Machine Learning Prediction of Multiple Infections in Elderly Surgery Patients | January 2012 - August 2018
  Utilizing machine learning techniques, investigators developed the geriatric infection assessment model, leveraging domestic databases to predict multiple postoperative infections in elderly patients.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, Study Chair — Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital
Locations (1):
- Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital, Beijing, Beijing Municipality, China